CLINICAL TRIAL: NCT07052890
Title: Role of a Food Supplement Containing Curcumin, Green Tea and Vitamin D on Symptom Control in Diarrhoea Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Curcumin, Vitamin D and Green Tea in IBS-D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Consultant Clinical Scientist, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FGC-24-002
Record Dates: First submitted 2025-06-10; First posted 2025-07-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome (IBS); Irritable Bowel Syndrome With Diarrhea (IBS-D)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Curcumin; Vitamin D; Tea

STUDY DESIGN:
Intervention Model Description: The study will utilise a double blind design with 1:1 active to placebo, with crossover to open label treatment. The study comprises of a 2 week screening period followed by a 4 week randomised treatment period. At the end of the randomisation treatment period, participants will all receive active treatment open label for a further 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 28 days placebo capsules 4x daily, followed by 28 days of open label active treatment
  Interventions: Dietary Supplement: Placebo Capsule(s)
- Curcumin, Vitamin D and Green tea (Experimental): 28 days Curcumin, Vitamin D and Green tea capsules 4x daily, followed by a further 28 days of this treatment but non-blinded (open label)
  Interventions: Dietary Supplement: Curcumin, vitamin d and green tea extract; Dietary Supplement: Placebo Capsule(s)

INTERVENTIONS:
Dietary Supplement: Curcumin, vitamin d and green tea extract — A combination of the following ingrediants per 4 capsules:
  CurcuWin® 1000mg - of which 200mg Curcuminoids
  Green Tea Extract 400mg - (0.1-0.5% caffeine)
  Vitamin D₃ 50 µg 2000IU
  Arms: Curcumin, Vitamin D and Green tea
Dietary Supplement: Placebo Capsule(s) — Placebo - identical capsules containing inert color matched power

SUMMARY:
Irritable Bowel Syndrome (IBS) is a highly prevalent condition of the gastrointestinal tract that has significant impact on sufferer's quality of life. The diarrhoea variant (IBS-D) makes up around one third of all IBS sufferers. There is currently a lack of both effective pharmacological and non-pharmacological treatments for IBS-D.

Three food supplements: Green tea, vitamin D and curcumin have all been shown to demonstrate benefit in either reducing symptoms in IBS or diarrhoea as individual ingredients, but have never been tested in combination to assess their effectiveness in IBS. This research study aims to examine the effectiveness of green tea, vitamin D and curcumin in combination compared to a placebo capsule in individual suffering from IBS-D.

The study will aim to enroll 78 participants with IBS-D and utilise a placebo-controlled double blind design. The study will consist of a 2 week screening period, a 4 week randomised treatment period (50% participants to receive placebo, 50% to receive active treatment), followed by a 4 week open label treatment period (all participants to receive the active study product).

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Participant has irritable bowel syndrome with diarrhoea (IBS-D), as defined by the Rome IV criteria.
3. Participant has an IBS-SSS score of >175 at screening.
4. Participant is a male or non-pregnant female and is ≥18 years of age
5. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.
6. Participant has capacity to understand written English.
7. Participant has a body mass index (BMI) of 18.5 - 39.9kg/m2 (bounds included).
8. Participant agrees to follow all pre-test preparation before breath testing visits.

Exclusion Criteria:

1. Prior abdominal surgery other than appendectomy and cholecystectomy.
2. Known hypercalcaemia.
3. Participating in another trial or taken an IMP within the last 1 month.
4. Females who report to be pregnant or lactating
5. Unwilling to maintain stable doses of permitted concomitant medication
6. Unwilling to maintain a stable diet for the duration of the trial
7. Being in the opinion of the investigator unsuitable
8. Insufficient knowledge of English to complete the daily bowel diary and food diary
9. Hypersensitivity to any component of the supplement
10. Hypersensitivity or known allergy to lactulose
11. Drug interactions with any component of the supplement
12. Consumption of antibiotics, prebiotics or probiotics (in food products or as supplements) in the last 4 weeks prior to, or during the study.
13. Vitamin D two week washout
14. Participants who have received bowel preparation for investigative procedures in the 4 weeks prior to the study
15. Individuals declaring additional specific dietary needs
16. Inflammatory bowel disease or coeliac disease
17. Any other condition, deemed by the investigator, that may be causing their symptoms
18. No major co-morbidity.
19. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or Sponsor member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean decrease of Irritable bowel syndrome symptom severity score (IBS-SSS) | From Enrollment to end of 4 week randomised treatment period
  Mean change in IBS-SSS at the end of the randomised treatment phase between Active and placebo arms.
  The IBS-SSS is numeric score based on 5 questions (each rated 0-100), with a total minimum score of 0 and maximum of 500, with a higher score indicating greater severity of symptoms.

SECONDARY OUTCOMES:
Use of rescue medication | 4 weeks
  Average change in rescue medication use from week 1 of randomisation period compared to week 4 of randomisation period, between active and placebo arms
Assessment of change breath methane levels during hydrogen and methane breath testing (HMBT) | 4 weeks
  Assessment of effect of active treatment vs placebo on breath hydrogen levels from baseline to end of randomised treatment period.
  Breath hydrogen levels will be measured using a lactulose hydrogen and methane breath test. Total area under the curve for methane during the test will be calculated.
Mean change irritable bowel syndrome quality of life (IBS-QoL) questionnaire score | 4 weeks
  Mean change IBS-QoL scores from baseline to end of randomised treatment period, between active and placebo groups.
  The IBS-QoL questionnaire is made up of 34 questions each scored 1-5. Higher scores indicate better quality of life. Lower scores suggest more severe impact of IBS on daily living.
Longevity of treatment effect | 8 weeks
  Longevity of treatment effect assessed in the active group with comparison of IBS-SSS scores from the randomised treatment period to end of open label period.
  The IBS-SSS is numeric score based on 5 questions (each rated 0-100), with a total minimum score of 0 and maximum of 500, with a higher score indicating greater severity of symptoms.
Stool Consistency | 4 weeks
  Stool Consistency assessed as average number of days with Bristol Stool Scale type (mean over 4 weeks, mean of first week and last week of the randomisation period).
  A favorable change in mean score would be changes from type 6 or 7 stools (diarrhoea type stool consistency) to type 3,4,5 stools, which are considered normal stool consistency.
Stool frequency | 4 weeks
  Stool Frequency (mean of 4 weeks, mean of first week and last week of the randomisation period)
Change in bloating measured using daily bowel diary. | 4 weeks
  Change in average daily bloating score for week 1 of the randomised treatment period to week 4 of the randomised treatment period.
  Severity of bloating will be scored daily by participants on a scale of 0-3, 0 being no bloating, 3 being severe bloating.
Change in abdominal pain measured using the daily bowel diary | 4 weeks
  Change in average daily abdominal pain score for week 1 of the randomised treatment period to week 4 of the randomised treatment period.
  Severity of abdominal pain will be scored daily by participants on a scale of 0-3, 0 being no bloating, 3 being severe bloating.
Breath Hydrogen levels measured using hydrogen and methane breath testing (HMBT) | 4 weeks
  Assessment of effect of active treatment vs placebo on breath hydrogen levels from baseline to end of randomised treatment period.
  Breath hydrogen levels will be measured using a lactulose hydrogen and methane breath test. Total area under the curve for hydrogen during the test will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, PhD, Principal Investigator — The Functional Gut Clinic
Locations (3):
- United Kingdom (3):
  - The Functional Gut Clinic Cambridge, Cambridge
  - The Functional Gut Clinic London, London
  - The Functional Gut Clinic Manchester, Manchester

IPD SHARING:
Plan to Share IPD: Undecided